CLINICAL TRIAL: NCT05725980
Title: A Retrospective Cephalometric Study on Upper Airways Changes Compared to Skeletal Angle Class and Divergence: a Retrospective Observational Study
Brief Title: Upper Airways Cephalometric Measures Compared to Skeletal Class and Divergence
Status: Completed | Type: Observational
Sponsor: Andrea Scribante (Other)
Responsible Party: Sponsor-Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Organization: University of Pavia (Other)
Other Study IDs: 2023-AIRWAYSCLASS
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Skeletal Malocclusion
Keywords: Upper airways dimensions; Skeletal Class; Skeletal Divergency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Skeletal Class I patients: Patients from this group present 0° < ANB < 4° on the cephalometric tracing.
  Interventions: Diagnostic Test: Cephalometric analysis
- Skeletal Class II patients: Patients from this group present ANB > 4° on the cephalometric tracing.
  Interventions: Diagnostic Test: Cephalometric analysis
- Skeletal Class III patients: Patients from this group present ANB < 0° on the cephalometric tracing.
  Interventions: Diagnostic Test: Cephalometric analysis

INTERVENTIONS:
Diagnostic Test: Cephalometric analysis — Cephalometric analysis will be performed evaluating upper airways landmarks.

SUMMARY:
The aim of the present study is to investigate the baseline upper airways dimensions in adult patients belonging to all skeletal classes

DETAILED DESCRIPTION:
Lateral cephalometric radiographs of adult orthodontic patients referring for orthodontic consultation at the Unit of Orthodontics and Pediatric Dentistry, Section of Dentistry, Department of Clinical, Surgical, Diagnostic and Pediatric Sciences, University of Pavia, 27100 Pavia, Italy, will be collected for the study according to the inclusion criteria.

For each lateral cephalometric radiograph, a cephalometric tracing will be performed with DeltaDent software (version 2.2.1, Outside Format, Spino d'Adda, Italy). Riedel's ANB angle [Riedel 1952] has been adopted to determine patients' skeletal class. Steiner's SN^GoGn angle [Steiner 1953] will be used to evaluate skeletal divergence. Biprotrusion will be assessed for SNA > 84° and SNB > 82°, while biretrusion for SNA < 80° and SNB < 78°.

Sample size calculation was performed with "soft palate length" as primary outcome. Considering alpha = 0.05 and power = 95%, an expected mean value of 31.05 with a standard deviation of 4.16 was hypothesized, with an expected mean difference of 3.34 [Sprenger et al. 2017], therefore 40 patients per group were required.

Statistical analysis will be conducted with R® software (version 3.1.3 R Development Core Team, R Foundation for Statistical Computing, Wein, Austria). For each cephalometric measure belonging to the three skeletal classes, descriptive statistics (mean and standard deviation) will be calculated. Appropriate statistical tests will be used to assess data normality and multiple comparisons. Linear regressions will be performed between upper airways diameters and SNA, SNB, ANB, SN^GoGn, ANSPNS^GoGn, PT, PL, sex and age.

ELIGIBILITY:
Inclusion Criteria:

* Patients with permanent dentition
* Caucasian patients
* Patients with one lateral cephalometric digital radiograph executed in Natural Head Position (patients were asked to keep the teeth in contact and the lips relaxed).

Exclusion Criteria:

* maxillo-facial traumas
* nasopharyngeal pathologies
* craniofacial dysmorphisms
* orthognatic surgery
* radiographs not performed in Natural Head Position
* unsuitable radiographs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients referring to the Unit of Orthodontics and Pediatric Dentistry for orthodontic consultation.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
NL (nasopharynx length) | Baseline
  Distance between Ad1 and PNS
PD (nasopharynx depth) | Baseline
  Line parallel to bispinal plane and connecting PNS and the posterior margin of pharynx
SPAS (Superior Pharyngeal Airway Space) | Baseline
  From the half of the posterior wall of soft palate (MMP) perpendicularly to the closest point on the posterior of the posterior wall of the pharynx
MAS (Mean Airway Space) | Baseline
  U1-U2 distance
PAS min (Pharyngeal Airway Space minimum) | Baseline
  T1-T2 distance along Go-B parallel line
IAS (Inferior Airway Space) | Baseline
  From the superior margin of the epiglottis (Ph1) to the closest perpendicular point on the posterior wall of the pharynx
LPW (Lateral Pharyngeal Wall) | Baseline
  Distance between epiglottic vallecula (Va1) and the posterior wall of pharynx perpendicular to Va1
PT | Baseline
  Soft palate thickness
PL | Baseline
  Soft palate length
MPH (Mandibular Plane - Hyoid bone) | Baseline
  Distance from the most anterior and superior point of the hyoid bone (H1) perpendicular to mandibular plane

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.